CLINICAL TRIAL: NCT04361708
Title: A Phase 1 Dose Finding Study of the gFOLFOXIRITAX Regimen Using UGT1A1 Genotype-directed Irinotecan With Fluorouracil, Leucovorin, Oxaliplatin and Taxotere in Patients With Untreated Advanced Upper Gastrointestinal Adenocarcinomas: The I-FLOAT Study
Brief Title: Safety of Combining Irinotecan With 5-FU, Leucovorin/Folinic Acid, Oxaliplatin, and Docetaxel Chemotherapies
Acronym: I-FLOAT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-1292
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Oxaliplatin; Docetaxel; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- High Risk UGT1A1 genotype (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil
- Intermediate Risk UGT1A1 genotype (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil
- Low Risk UGT1A1 genotype (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered on day 1 of each cycle at 85mg/kg. The drugs will be given through the patient's Mediport. It will be given once every 14 days (2 weeks), on days 1 and will be continued for 8 doses (4 months)
Drug: Docetaxel — Docetaxel will be administered on day 1 of each cycle at 25mg at dose level 1; 37.5 at dose level 2. The drugs will be given through the patient's Mediport.It will be given once every 14 days (2 weeks), on days 1 and will be continued for 8 doses (4 months)
Drug: Leucovorin — Leucovorin will be administered on day 1 of each cycle at 400mg/kg. The drugs will be given through the patient's Mediport. It will be given once every 14 days (2 weeks), on days 1 and will be continued for 8 doses (4 months)
Drug: Irinotecan — Irinotecan will be administered on day 1 of each cycle at 120mg/m2 for low risk group, 105mg/m2 for intermediate risk group, 45mg/m2 for high risk group . The drugs will be given through the patient's Mediport. It will be given once every 14 days (2 weeks), on days 1 and will be continued for 8 doses (4 months)
Drug: 5-Fluorouracil — 5-FU is given as a continuous intravenous infusion over 2 days. Patient can receive the 2-day infusion as an outpatient. On day 3 of each cycle, the patient will return to the infusion center to have the infusion hook-up disconnected.

SUMMARY:
The purpose of the proposed study is to establish the safety of combining irinotecan chemotherapy with 5-FU, leucovorin/folinic acid, oxaliplatin, and docetaxel (abbreviated as the I-FLOAT study of gFOLFOXIRITAX) chemotherapies (leucovorin/folinic acid is a vitamin to make 5-FU work well).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic pancreatic adenocarcinoma, gastroesophageal adenocarcinoma, cholangiocarcinoma, gallbladder adenocarcinoma, ampullary carcinoma, adenocarcinoma of unclear primary (with upper GI primary suspected), or other primary GI malignancy for which the treating physician feels that I-FLOAT is a reasonable therapeutic option.
2. Patients with a history of obstructive jaundice due to the primary tumor must have resolved to <1.5 X upper limit of normal and a metal biliary stent in place
3. Age greater than or equal to 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status =1
5. Life expectancy > 3 months
6. Adequate organ function, as defined by each of the following:

   Absolute neutrophil count (ANC) = 1500/uL Hemoglobin > 9g/dL (transfusion permitted with stability for > 1 week) Platelets > 100,000/uL Total bilirubin = 1.5 mg/dL AST and ALT = 2.5 X upper limit of normal; alkaline phosphatase = 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis.

   AST and ALT = 5 X upper limit of normal if hepatic metastases are present. Creatinine = 1.5 mg/dL
7. Measurable or non-measurable disease will be allowed.
8. Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment.
9. Negative serum or urine B-hCG pregnancy test at screening for patients of childbearing potential
10. Patients taking substrates, inhibitors, or inducers of CYP3A4 should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with irinotecan.

Exclusion Criteria:

1. Prior radiation therapy for any cancer.
2. Prior chemotherapy for metastatic disease Recurrence of disease within 6 months of perioperative chemotherapy are eligible if other eligibility criteria are met
3. Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
4. Diarrhea, grade 1 or greater by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v. 4.0*). Pancreatic cancer patients with clinical evidence of pancreatic insufficiency must be taking pancreatic enzyme replacement.
5. Neuropathy, grade 2 or greater by NCI-CTCAE, v. 4.0.
6. Documented brain metastases
7. Serious underlying medical or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment.
8. Active uncontrolled bleeding.
9. Pregnancy or breastfeeding.
10. Major surgery within 4 weeks.
11. Previous or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer for which the patient has been previously treated and the lifetime recurrence risk is less than 30%, and meets all other eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The maximum dose tolerated | 1 month
  To determine the maximum tolerated dose in the first month of therapy in each of the three main genotype groups (low, intermediate, and high risk) using genotype-guided dosing of irinotecan as part of the I-FLOAT regimen

SECONDARY OUTCOMES:
Cumulative dose of each chemotherapy drug | 4 months
  To determine the cumulative dose of each chemotherapy drug (irinotecan, 5-FU, oxaliplatin, docetaxel) administered in each genotype group over a period of 4 months (8 doses).
Total duration of therapy | 18 months
  To determine the total duration of therapy, which would be administered perioperatively in future studies for the curative-intent setting.
Overall Response Rate | 5 years
  To determine early efficacy (overall responsive rate, progression free survival, and overall survival) in all patients enrolled and treated in the study.
Progression free survival rate | 5 years
  To determine early efficacy (overall responsive rate, progression free survival, and overall survival) in all patients enrolled and treated in the study.
Overall survival rate | 5 years
  To determine early efficacy (overall responsive rate, progression free survival, and overall survival) in all patients enrolled and treated in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catenacci, MD, Principal Investigator — University of Chicago Medicine
Locations (1):
- The University of Chicago, Chicago, Illinois, United States